CLINICAL TRIAL: NCT05668338
Title: MED-EL HEARING SOLUTIONS (MEHS): AN OBSERVATIONAL STUDY
Acronym: MEHS
Status: Recruiting | Type: Observational
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: MED-EL_CRD_2015_06
Record Dates: First submitted 2022-12-05; First posted 2022-12-29 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Implantable or non-implantable MED-EL hearing solution — Receipt of an implantable or non-implantable MED-EL hearing solution

SUMMARY:
This Registry represents a non-interventional systematic collection of clinical data in which prospective data from children and adults are collected as fully anonymized data sets, derived from original clinical records on appropriately informed subjects.

This is a patient-outcomes Registry for subjects of any age who are provided in routine clinical practice with one or more MED-EL hearing devices. The Registry aims to collect data for hypothesis generation on subject device use, auditory performance, quality of life and health-related utilities, across different types of implantable and non-implantable hearing devices from MED-EL company. Subjects will be evaluated with a set of standardized tests and questionnaires prior to implantation or prior to initial device activation (baseline) and at follow-up intervals according to the clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* For children and adults receiving an implant: Subjects submitted or planned to be submitted to unilateral or bilateral implantation, using simultaneous or sequential procedures.
* For children and adults receiving a non-implantable device: Subjects submitted or planned to be submitted to unilateral or bilateral treatment with a non-implantable device from MED-EL.
* Unilateral, bilateral or bimodal users (children and adults) of cochlear implants (CIs), electric-acoustic devices, bone conduction implants, middle ear implants or any other implantable or non-implantable hearing solution from MED-EL.
* Signed written informed consent for data collection for Registry purposes.

Exclusion Criteria:

* Lack of compliance with any inclusion criteria.
* Anything that, in the opinion of the Investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the Registry procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: No study population defined
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-06-26 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Subject Demographics | 5 years
Hearing Threshold level | 5 years
  Audiometry testing (unaided)
Speech test | 5 years
  Results from speech tests
HISQUI (Hearing Implant Sound Quality Index) | 5 years
  Results from the HISQUI questionnaire
APHAB (Abbreviated Profile of Hearing Aid Benefit) | 5 years
  Results from the APHAB questionnaire
ASC (Auditory Skills Checklist) | 5 years
  Results from the ASC questionnaire
APSQ (Audio Processor Satisfaction Questionnaire) | 5 years
  Results from the APSQ questionnaire
LEAQ (LittlEars Auditory Questionnaire) | 5 years
  Results from the LEAQ questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Müller, Prof.Dr.med, Principal Investigator — Klinikum der Universität München Campus Großhadern
Locations (8):
- Germany (8):
  - Katholisches Klinikum Bochum, Bochum
  - Universitätsklinik Carl Gustav Carus - Klinik und Poliklinik für Hals-, Nasen- und Ohrenheilkunde, Dresden
  - Universitätsklinikum der Goethe-Universität, Frankfurt
  - Sektion Otologie und Neuro-Otologie UNI-Klinikum Heidelberg, Heidelberg
  - Klinikum der Universität München Campus Großhadern, München
  - Evangelisches Krankenhaus Oldenburg, Oldenburg
  - Klinik und Poliklinik für Hals-, Nasen-, Ohrenheilkunde, Kopf- und Halschirurgie "Otto Körner", Rostock
  - Universitätsklinikum Tübingen, Klinik für Hals-, Nasen- u. Ohrenheilkunde, Plastische Operationen, Tübingen

IPD SHARING:
Plan to Share IPD: No